CLINICAL TRIAL: NCT00001416
Title: Skeletal Responses to Macrophage-Targeted Glucocerebrosidase in Patients With Type 1 Gaucher's Disease
Brief Title: Bone Response to Enzyme Replacement in Gaucher's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 940050; 94-N-0050
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Gaucher's Disease
Keywords: Bone Disease; Calcitriol; Enzyme Replacement Therapy; Gaucher's Disease; Vitamin D
MeSH Terms: conditions — Gaucher Disease; Bone Diseases | interventions — alglucerase

INTERVENTIONS:
Drug: CEREDASE™

SUMMARY:
The purpose of this study is to examine how the skeleton responds to repeated doses of enzyme replacement therapy in patients with type I Gaucher's disease who have had their spleens removed.

Gaucher disease is a lysosomal storage disease resulting from glycocerebroside accumulation in macrophages due to a genetic deficiency of the enzyme glucocerebrosidase. It may occur in adults but occurs most severely in infants, in whom cerebroside also accumulates in neurons. Patients with Gaucher's disease experience enlargement of the liver and spleen and bone destruction. The condition is passed from generation to generation through autosomal recessive inheritance.

Type I is the most common form. It is a chronic non-neuronopathic form, meaning the disease does not affect nerve cells. The symptoms of type I can appear at any age.

In this study patients will be divided into three groups. Each group will receive different doses of enzyme replacement (Ceredase). In addition, two of the three groups will also receive doses of a form of vitamin D (calcitriol). Researchers believe the groups receiving vitamin D will have an improved response as compared to those patients only receiving enzyme replacement.

Patients in each group who respond to enzyme replacement with increases in bone density will be compared to the other treatment groups.

DETAILED DESCRIPTION:
The purpose of this study is to examine the response of the skeleton to repeated infusions of macrophage-targeted glucocerebrosidase (CEREDASE (Trademark) ) in splenectomized patients with type I Gaucher's disease. The magnitude and rate of development of the skeletal response will be monitored non-invasively. Theoretically, an enhanced response should occur in patients supplemented with pharmacologic doses of 1, 25-dihydroxyvitamin D3 (calcitriol), since calcium absorption and enzyme delivery to bone marrow macrophages should be increased in this setting. These issues will be addressed in a clinical trial that uses a modified factorial design. A total of 57 patients will be assigned to three treatment groups by block randomization.

Group 1: CEREDASE (Trademark) (60 IU/kg q2wks; 0-6 months)

CEREDASE (Trademark) (30 IU/kg q2wks; 7-24 months)

Group 2: Calcitriol (0.25-3.0 micrograms/day; 0-24 months)

CEREDASE (Trademark) (60 IU/kg q2wks; 7-12 months)

CEREDASE (Trademark) (30 IU/kg q2wks; 13-24 months)

Group 3: Calcitriol (0.25-3.0 micrograms/day; 0-24 months)

CEREDASE (Trademark) (60 IU/kg q2wks; 0-6 months)

CEREDASE (Trademark) (30 IU/kg q2wks; 7-24 months)

The number of patients responding to enzyme replacement with a significant decrease in hepatic volume and a significant increase in trabecular bone density of the lumbar spine will be compared between the treatment groups.

ELIGIBILITY:
Splenectomized Gaucher patients.

Aged 18-45 who have not received enzyme therapy for at least 1 year.

No patients with other illnesses (pulmonary, liver, kidney, bone, hematologic).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1993-12; Study Completion 2000-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenthal DI, Barton NW, McKusick KA, Rosen BR, Hill SC, Castronovo FP, Brady RO, Doppelt SH, Mankin HJ. Quantitative imaging of Gaucher disease. Radiology. 1992 Dec;185(3):841-5. doi: 10.1148/radiology.185.3.1438773.
- [Background] Barton NW, Brady RO, Dambrosia JM, Di Bisceglie AM, Doppelt SH, Hill SC, Mankin HJ, Murray GJ, Parker RI, Argoff CE, et al. Replacement therapy for inherited enzyme deficiency--macrophage-targeted glucocerebrosidase for Gaucher's disease. N Engl J Med. 1991 May 23;324(21):1464-70. doi: 10.1056/NEJM199105233242104. PMID 2023606